CLINICAL TRIAL: NCT00011167
Title: Retinal Arteriolar Abnormalities and CV Mortality
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000-112; R01HL066018 (NIH); 960 (Other: Study Team)
Record Dates: First submitted 2001-02-13; First posted 2001-02-13 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Disorders; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cerebrovascular Disorders; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine whether retinal arteriolar changes (generalized narrowing, focal narrowing and arterio-venous nicking) and retinopathy were associated with 10-year stroke-and ischemic heart disease-related mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Blood vessels in the retina of the eye provide a valuable window for evaluating quantitatively small vessel arteriosclerosis (arteriolar narrowing, arterio-venous nicking and arterio-to-venule ratio (AVR)). Previous studies have suggested that these optic fundi vascular parameters may be useful measures of generalized vascular disease and may have important prognostic implications. This study addressed this issue in a quantitative way using an established cohort with previously acquired fundic photographs. The study addressed an important public health problem with findings that may identify at-risk patients who would benefit from earlier intervention.

The established cohort was from the Beaver Dam Eye Study cohort, a well-characterized population of predominantly white persons aged 43-86 years at the baseline in 1988-1990. The cohort was originally evaluated in 1988-1990 with routine clinical and laboratory evaluation plus high-quality optic fundi photos. The population had been followed over a 10-year period with identified deaths from ischemic heart disease or stroke.

DESIGN NARRATIVE:

This was a population-based case-cohort study to determine whether retinal arteriolar changes (generalized narrowing, focal narrowing and arterio-venous nicking) and retinopathy were associated with 10-year stroke-and ischemic heart disease-related mortality. The study population was selected from participants of the Beaver Dam Eye Study, a well-characterized population of predominantly white persons aged 43-86 years at the baseline examination in 1988-90. Cases were defined as participants who had died from either stroke or ischemic heart disease since the baseline examination. Three participants per case were selected from the cohort at baseline as controls, matched on gender and 5-year age intervals to cases. Focal arteriolar narrowing, arteriovenous nicking and retinopathy were graded to baseline using a standardized photographic grading protocol. To evaluate generalized arteriolar narrowing, a method modified from the Atherosclerosis Risk in Communities study was used. Retinal photographs were digitized and processed using a high-resolution scanner. Retinal arteriole and venule widths were then measured with the help of a computer program based on pixel density contrast between the vessel and the background retina. Finally, the average width of the arterioles was summarized as a retinal arteriole to venule ratio (AVR). Standard case-control methodology were applied to calculate the relative odds of association between generalized retinal arteriolar narrowing (using different categories of AVR) and other changes with stroke-and ischemic heart disease-related mortality. Logistic regression models controlling for potential confounders (e.g., blood pressure, serum lipid levels) were employed to evaluate the independent association between retinal arteriolar characteristics and stroke- and ischemic heart disease mortality.

ELIGIBILITY:
* Participated in the baseline examination of the Beaver Dam Eye Study in 1988-1990
* Had gradable fundus photographs taken at the baseline examination of the Beaver Dam Eye Study in 1988-1990

Ages: 43 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Beaver Dam Eye Study cohort was first identified by a private census of the city of Beaver Dam, Wisconsin from September 15, 1987 to May 4, 1988, was examined from 1988-90 (baseline examination), and re-examined in 1993-95 and 1998-2000. The baseline examination formed the population for both cases and controls. Cases were defined as study participants who had died since the baseline examination from stroke or ischemic heart disease. Three participants per case were selected from the entire cohort at baseline as controls, age and sex matched to cases, irrespective of vital status. No participants were recruited specifically for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1380 (Actual)
Dates: Start 2001-03; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Death due to stroke or ischemic heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Klein, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- [Background] Wong TY, Klein R, Nieto FJ, Klein BE, Sharrett AR, Meuer SM, Hubbard LD, Tielsch JM. Retinal microvascular abnormalities and 10-year cardiovascular mortality: a population-based case-control study. Ophthalmology. 2003 May;110(5):933-40. doi: 10.1016/S0161-6420(03)00084-8. PMID 12750093
- [Background] Knudtson MD, Klein BE, Klein R, Wong TY, Hubbard LD, Lee KE, Meuer SM, Bulla CP. Variation associated with measurement of retinal vessel diameters at different points in the pulse cycle. Br J Ophthalmol. 2004 Jan;88(1):57-61. doi: 10.1136/bjo.88.1.57. PMID 14693774
- [Background] Wong TY, Klein R, Klein BE, Meuer SM, Hubbard LD. Retinal vessel diameters and their associations with age and blood pressure. Invest Ophthalmol Vis Sci. 2003 Nov;44(11):4644-50. doi: 10.1167/iovs.03-0079. PMID 14578380
- [Background] Wong TY, Shankar A, Klein R, Klein BE, Hubbard LD. Retinal arteriolar narrowing, hypertension, and subsequent risk of diabetes mellitus. Arch Intern Med. 2005 May 9;165(9):1060-5. doi: 10.1001/archinte.165.9.1060. PMID 15883247
- [Background] Wong TY, Knudtson MD, Klein R, Klein BE, Meuer SM, Hubbard LD. Computer-assisted measurement of retinal vessel diameters in the Beaver Dam Eye Study: methodology, correlation between eyes, and effect of refractive errors. Ophthalmology. 2004 Jun;111(6):1183-90. doi: 10.1016/j.ophtha.2003.09.039. PMID 15177969
- [Background] Wong TY, Shankar A, Klein R, Klein BE, Hubbard LD. Prospective cohort study of retinal vessel diameters and risk of hypertension. BMJ. 2004 Jul 10;329(7457):79. doi: 10.1136/bmj.38124.682523.55. Epub 2004 Jun 2. PMID 15175230
- [Background] Wong TY, Knudtson MD, Klein R, Klein BE, Hubbard LD. A prospective cohort study of retinal arteriolar narrowing and mortality. Am J Epidemiol. 2004 May 1;159(9):819-25. doi: 10.1093/aje/kwh119. PMID 15105174
- [Background] Knudtson MD, Lee KE, Hubbard LD, Wong TY, Klein R, Klein BE. Revised formulas for summarizing retinal vessel diameters. Curr Eye Res. 2003 Sep;27(3):143-9. doi: 10.1076/ceyr.27.3.143.16049. PMID 14562179